CLINICAL TRIAL: NCT07321717
Title: A Randomized Controlled Trial Comparing The Analgesic Effectiveness Of Sacral Erector Spinae Plane Block And Penile Block In Children Undergoing Circumcision Surgery
Brief Title: Sacral Erector Spinae Plane Block Versus Penile Block For Analgesia In Pediatric Circumcision
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Münevver Kayhan, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ctf-sakral sünnet-03
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Sacral Erector Spinae Plane Block; Pediatric Regional Anesthesia; Regional Anaesthesia
Keywords: pediatric regional anesthesia; sacral ESP

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two independent groups: the Penile Nerve Block (PNB) group or the Sacral Erector Spinae Plane Block (sacral ESPB) group. Each participant will receive only the assigned intervention and will be followed throughout the perioperative and postoperative period. The parallel design allows comparison of analgesic effectiveness, safety, and postoperative outcomes between the two independent groups
Who Masked: Participant, Outcomes Assessor
Masking Description: This study is double-blind to compare the analgesic effectiveness and safety of Penile Nerve Block (PNB) and Sacral Erector Spinae Plane Block (sacral ESPB) in pediatric circumcision. Participants (children) and outcome assessors are unaware of group assignment to minimize bias. Postoperative pain and outcomes are measured using the FLACC scale (Face, Legs, Activity, Cry, Consolability), where higher scores indicate more severe pain and lower scores less pain. Only the anesthesiologists performing the blocks know the assigned intervention for safety and correct technique; they do not collect postoperative data. Blinding ensures objective assessment of pain, analgesic consumption, hemodynamic changes, and complications during the perioperative and postoperative period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Penile Nerve Block (PNB) group (Active Comparator): Participants in this group will receive the standard penile nerve block prior to surgery. The block is performed by subcutaneous infiltration of 0.5 ml/kg of 0.25% bupivacaine around the ventral penoscrotal junction and base of the penis. This is the standard clinical practice group used for comparison.
  Interventions: Procedure: Penile Nerve Block (PNB)
- Sacral Erector Spinae Plane Block (SESPB) group (Experimental): Participants in this group will receive a sacral ESPB before circumcision surgery. The block is performed with 0.5 ml/kg of 0.25% bupivacaine under ultrasound guidance using an in-plane, craniocaudal approach while the child is in the prone position. This is the investigational intervention being studied for analgesic effectiveness and safety.
  Interventions: Procedure: Sacral Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Sacral Erector Spinae Plane Block — Participants will receive a sacral ESPB prior to circumcision surgery. 0.5 ml/kg of 0.25% bupivacaine is injected under ultrasound guidance using an in-plane, craniocaudal approach while the child is in the prone position. This is the investigational procedure being studied for analgesic effectiveness and safety.
  Arms: Sacral Erector Spinae Plane Block (SESPB) group
Procedure: Penile Nerve Block (PNB) — Participants will receive the standard penile nerve block prior to surgery. 0.5 ml/kg of 0.25% bupivacaine is infiltrated subcutaneously around the ventral penoscrotal junction and base of the penis. This serves as the standard comparator.
  Arms: Penile Nerve Block (PNB) group

SUMMARY:
Circumcision is one of the most frequently performed surgical procedures in childhood and is associated with significant postoperative pain. This randomized controlled trial (RCT) aims to compare the analgesic effectiveness of sacral erector spinae plane block (sacral ESPB) and penile nerve block (PNB) in children undergoing circumcision surgery. The primary outcome is postoperative pain, assessed using the Face, Legs, Activity, Cry, and Consolability (FLACC) scale at predefined time intervals within the first 24 hours after surgery. Secondary outcomes include intraoperative analgesic consumption, time to first postoperative analgesic requirement, perioperative hemodynamic changes. The results of this study are expected to provide evidence for selecting the optimal regional analgesic technique for pediatric circumcision surgery.

DETAILED DESCRIPTION:
Circumcision is one of the most commonly performed surgical procedures in childhood and is associated with significant postoperative pain. Inadequate analgesia in pediatric patients may lead to adverse hemodynamic, hormonal, metabolic, and immunological responses, as well as increased agitation and discomfort. Therefore, a multimodal analgesia (MMA) approach is recommended to prevent the onset of pain and provide effective perioperative analgesia. Regional anesthesia (RA) techniques offer safe, effective, and hemodynamically stable analgesia in pediatric patients. Penile nerve block (PNB) is a commonly used RA technique for circumcision, performed by subcutaneous infiltration of local anesthetic around the glans penis and penoscrotal junction. More recently, the sacral erector spinae plane block (sacral ESPB) has been introduced as an alternative RA method, providing wide analgesic coverage by affecting the pudendal nerve and its branches. Sacral ESPB has been successfully applied in pediatric urogenital and anorectal surgeries, demonstrating effective postoperative analgesia.

This randomized controlled trial (RCT) aims to compare the analgesic effectiveness of sacral ESPB and PNB in children aged 1-12 years with American Society of Anesthesiologists (ASA) physical status I-II undergoing circumcision surgery. Participants will be randomly allocated using a closed-envelope method to one of two groups. The PNB group will receive 0.5 mL/kg of 0.25% bupivacaine via circumferential subcutaneous injection along the penoscrotal line. The sacral ESPB group will receive 0.5 mL/kg of 0.25% bupivacaine under ultrasound (USG) guidance using an in-plane, cranio-caudal technique. All procedures will be performed by pediatric anesthesia faculty experienced in RA. Premedication will include intravenous (IV) midazolam 0.05 mg/kg and ketamine 0.5 mg/kg. General anesthesia (GA) will be induced with IV propofol 2-3 mg/kg, fentanyl 1 µg/kg, and rocuronium 0.6 mg/kg, followed by endotracheal intubation and maintenance with sevoflurane 1 minimum alveolar concentration (MAC). Intraoperative monitoring will include electrocardiography (ECG), peripheral oxygen saturation (SpO₂), and non-invasive blood pressure (NIBP). Hemodynamic changes exceeding 20% from baseline will be treated with remifentanil infusion.

Blinding (Körleme): This study will be conducted using a double-blind design. The patients and the investigators responsible for postoperative pain assessment and data collection will be unaware of group allocation. Only the anesthesiologists performing the blocks will know which intervention (PNB or sacral ESPB) is administered to ensure patient safety. This approach minimizes bias and ensures objective evaluation of outcomes.

Postoperative pain will be assessed using the Face, Legs, Activity, Cry, and Consolability (FLACC) scale, which ranges from 0 to 10 points. A higher FLACC score indicates more severe pain, while a lower score indicates less pain. Analgesic administration will follow a standardized protocol: FLACC ≤3 indicates sufficient analgesia; FLACC 4-6 will be treated with IV paracetamol 10 mg/kg; FLACC ≥7 will be treated with IV fentanyl 0.5 µg/kg in the recovery unit. On the ward, oral paracetamol 10 mg/kg or ibuprofen 10 mg/kg will be administered according to FLACC scores. Phone follow-up at 16 and 24 hours will monitor pain scores and rescue analgesic consumption.

The primary outcome is postoperative pain within the first 24 hours as measured by FLACC scores. Secondary outcomes include intraoperative analgesic consumption, time to first postoperative analgesic requirement, perioperative hemodynamic changes, time to first urination, parental satisfaction, and postoperative adverse events such as nausea, vomiting, or block-related complications.

This study aims to determine the optimal regional analgesic technique for pediatric circumcision surgery by comparing the efficacy, safety, and satisfaction outcomes of sacral ESPB and PNB.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 and 12 years
* Scheduled for circumcision surgery
* Classified as American Society of Anesthesiologists (ASA) physical status I-II
* Written informed consent obtained from both the participant (when appropriate) and their parents or legal guardians

Exclusion Criteria:

* Age under 1 year or over 12 years
* Undergoing circumcision combined with other surgical procedures
* Presence of neurological deficits
* History of bleeding diathesis
* Allergy to local anesthetic (LA) drugs
* Redness or infection at the injection site
* Presence of congenital sacral anomalies
* Mental retardation
* Psychiatric disorders or kidney disease
* Refusal to participate in the study

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Scores within 24 Hours | 0-24 hours after circumcision surgery
  Postoperative pain will be assessed using the FLACC scale (Face, Legs, Activity, Cry, Consolability) at multiple time points (0, 1, 2, 4, 8, 12, 16, and 24 hours postoperatively). Scores range from 0-10, where higher scores indicate more severe pain and lower scores indicate less pain. The primary outcome is the comparison of pain levels between the Sacral Erector Spinae Plane Block (SESPB) group and the Penile Nerve Block (PNB) group during the first 24 hours after surgery.

SECONDARY OUTCOMES:
Total Analgesic Consumption in 24 Hours | 0-24 hours postoperatively
  Total amount of analgesics (intravenous and oral) administered within the first 24 hours after surgery will be recorded.
Intraoperative Analgesic Consumption | During surgery
  Total dose of remifentanil administered intraoperatively will be recorded and compared between the SESPB and PNB groups.
Time to First Analgesic Requirement | 0-24 hours postoperatively
  Time from the end of surgery to the first need for rescue analgesia will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Munevver Kayhan, Principal Investigator — Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty; Pinar Kendigelen, Study Chair — Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty; Ayse Cigdem Tutuncu, Professor Doctor, Study Chair — Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty; Ali Ekber Hakalmaz, Lecturer Doctor, Study Chair — Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty
Locations (1):
- Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty, Bakırköy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No